CLINICAL TRIAL: NCT02756273
Title: Impact of a Bridge Device on the Loop Ileostomy
Acronym: IBIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier de Beauvais (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2015_843_0008; 2015-A00620-49 (Other: ANSM); 2015/29 (Other: CPP Nord Ouest II)
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Elective Colorectal Surgery
Keywords: ileostomy; morbidity; colorectal surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- no bridge device (Experimental): After the ileostomy creation, no bridge device was placed.
  Interventions: Device: no bridge device
- bridge device (Active Comparator): A bridge device was placed after the stoma creation.
  Interventions: Device: bridge device

INTERVENTIONS:
Device: bridge device
  Arms: bridge device
Device: no bridge device
  Arms: no bridge device

SUMMARY:
During the creation of an ileostomy, a bridge device is systematically placed in an aim to reduce wound and peritoneal contamination by stools. Nevertheless no evidence was reported to justify this issue.

Moreover the placement of a bridge device increases the difficulty of nurse cares and is associated with its own morbidity.

ELIGIBILITY:
Inclusion Criteria:

* colorectal disease (cancer; diverticulitis; Crohn disease; inflammatory bowel disease)
* requiring elective surgery with an ileostomy
* patient having given his consent before the enrollment

Exclusion Criteria:

* patient with early closure of the stoma (within 10 days after the colorectal surgery)
* long term corticoids
* emergency surgery
* history of stoma in the side of the stoma placement planned for the study
* BMI >50
* No signature of the consent to participate in the study
* Physical or mental state not allowing participation in the study
* Contraindication to surgery
* ASA classification (American Society of Anesthesiologists) IV-V or life expectancy <48h
* Pregnancy or breastfeeding
* Patient under guardianship or guardianship or patient deprived of liberty by a judicial or administrative decision (in accordance with articles L1121-6 and L1121-8 of the Public Health Code)
* Minor patient
* Patient without social protection

Peroperative exclusion criteria:

* no anastomosis
* no ileostomy
* Spontaneous stomal retraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-10-02 (Estimated)

PRIMARY OUTCOMES:
absence of postoperative morbidity | two months after the surgery
  the primary outcome is a composite score. The complication is considered as present if the patient experienced at least one of the following events: surgical site infection (either superficial, deep or distant); a parastomal irritation; a stomal necrosis; parastomal hernia; a stoma stenosis; a stoma prolapsus or a stoma leakage. The primary endpoint is evaluated by a nurse devoted to stoma care according to an open label.

SECONDARY OUTCOMES:
difficulty of the stoma conception | at the end of the surgery
  the difficulty was assessed by the surgeon thanks to a score ranging from 1 to 10.
the reoperation rate | postoperative month one
  the reoperation rate is defined as the number of reoperation one month after the colorectal surgery
the mortality rate | postoperative month one
  the mortality rate is defined as the number of deaths one month after the surgery
the postoperative morbidity | postoperative month one
  the postoperative morbidity is defined according the Clavien - Dindo classification and corresponds to the number of patients with a postoperative outcome
the specific quality of life | postoperative year one
  the quality of life is assessed with the STOMA QoL form at Baseline, 2, 6 months after the surgery and one year after the surgery
the rate of stoma closure | 6 months after the surgical procedure
  the rate of stoma closure is defined as the number of patients for whom the stoma was closed 6 months after the colorectal surgery.
the rate of anastomotic fistula | 2 months after the colorectal surgery
  the rate of anastomotic fistula is defined as the number of anastomotic fistula after the colorectal surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Charles SABBAGH, Principal Investigator — CHU Amiens Picardie
Locations (3):
- France (3):
  - Amiens Universitary Hospital, Amiens
  - Beauvais hospital, Beauvais
  - Chu Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matthiessen P, Hallbook O, Rutegard J, Simert G, Sjodahl R. Defunctioning stoma reduces symptomatic anastomotic leakage after low anterior resection of the rectum for cancer: a randomized multicenter trial. Ann Surg. 2007 Aug;246(2):207-14. doi: 10.1097/SLA.0b013e3180603024. PMID 17667498
- [Background] Sagap I, Remzi FH, Hammel JP, Fazio VW. Factors associated with failure in managing pelvic sepsis after ileal pouch-anal anastomosis (IPAA)--a multivariate analysis. Surgery. 2006 Oct;140(4):691-703; discussion 703-4. doi: 10.1016/j.surg.2006.07.015. PMID 17011918
- [Background] Panis Y, Maggiori L, Caranhac G, Bretagnol F, Vicaut E. Mortality after colorectal cancer surgery: a French survey of more than 84,000 patients. Ann Surg. 2011 Nov;254(5):738-43; discussion 743-4. doi: 10.1097/SLA.0b013e31823604ac. PMID 21997816
- [Background] Oberkofler CE, Rickenbacher A, Raptis DA, Lehmann K, Villiger P, Buchli C, Grieder F, Gelpke H, Decurtins M, Tempia-Caliera AA, Demartines N, Hahnloser D, Clavien PA, Breitenstein S. A multicenter randomized clinical trial of primary anastomosis or Hartmann's procedure for perforated left colonic diverticulitis with purulent or fecal peritonitis. Ann Surg. 2012 Nov;256(5):819-26; discussion 826-7. doi: 10.1097/SLA.0b013e31827324ba. PMID 23095627
- [Background] Cottam J, Richards K, Hasted A, Blackman A. Results of a nationwide prospective audit of stoma complications within 3 weeks of surgery. Colorectal Dis. 2007 Nov;9(9):834-8. doi: 10.1111/j.1463-1318.2007.01213.x. Epub 2007 Aug 2. PMID 17672873
- [Derived] Sabbagh C, Mauvais F, Demouron M, Browet F, Tartar L, Hariz H, Bridoux V, Tuech JJ, Diouf M, Regimbeau JM. Is a bridge (rod) necessary for loop ileostomy? A phase II randomized control trial. Tech Coloproctol. 2025 Mar 25;29(1):87. doi: 10.1007/s10151-025-03132-4. PMID 40131588